CLINICAL TRIAL: NCT05633225
Title: Measuring Central Sensitization and Physical Activity in Adolescents With Hypermobility Spectrum Disorder or Hypermobile Ehlers-Danlos Syndrome
Brief Title: Central Sensitization and Physical Activity in Adolescents With HSD/hEDS
Status: Completed | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Göteborg University (Other)
Responsible Party: Principal Investigator, Elke Schubert Hjalmarsson, RPT, Head of the occupational therapy and physiotherapy unit for children, Vastra Gotaland Region
Other Study IDs: CSaPhA-HSD/hEDS
Record Dates: First submitted 2022-10-19; First posted 2022-12-01 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Joint Hypermobility Syndrome; Hypermobile Ehlers-Danlos Syndrome
Keywords: Pain; Hypermobility; Physical activity; Central sensitization; Fatigue; Ehlers Danlos Syndrome
MeSH Terms: conditions — Ehlers-Danlos syndrome type 3; Pain; Motor Activity; Fatigue; Ehlers-Danlos Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient-group: Ninety adolescents, 13-17 years of age Diagnosed with Hypermobility Spectrum Disorder or hypermobile Ehlers Danlos Syndrome.
  Interventions: Other: Submax exercise test on a bicycle ergometer
- Control-group: Ninety adolescents, 13-17 years of age. Participants have to be pain free at time of investigation (NRS score <3/10)
  Interventions: Other: Submax exercise test on a bicycle ergometer

INTERVENTIONS:
Other: Submax exercise test on a bicycle ergometer — To achieve exertion and not exhaustion, cycling will be stopped at 75% of the expected maximum heart rate (maximum heart rate of 220 beats per minute minus age) as a target value.
  If the participant then indicated that they do not feel strained, the cycling will continue until the participant experienced an effort on Borg Rating of Perceived Exertion Scale scale of 15 (hard).

SUMMARY:
Hypermobility Spectrum Disorder and hypermobile Ehlers-Danlos Syndrome (HSD/hEDS) is under-recognized and poorly understood and its management is therefore not clear.

The goal of this study is to better understand pain and its impact on function in the daily activities of adolescents with Hypermobility Spectrum Disorder and/or hypermobile Ehlers-Danlos Syndrome.

This study will explore the presence of the pain sensitivity status after physical exercise as well as movement behaviour in adolescents with HSD/hEDS compared to a healthy control group.

DETAILED DESCRIPTION:
All participants will be asked not to undertake physical exercise at least 48 hours before the measurements, and to refrain from consuming caffeine, alcohol or nicotine. For ethical reasons, the patients are allowed to take non-opioid pain medicine as described in the first step of the World Health Organization analgesic ladder (COX-inhibitors and paracetamol), however the patients will be asked to abstain from these medications during the 24 hours period before the measurements.

ELIGIBILITY:
Inclusion criteria for the HSD/hEDS group:

* Able to read and understand Swedish
* Diagnosed with HSD or hEDS

Exclusion criteria for the HSD/hEDS group:

* Pregnancy and one year postpartum.
* Other syndromes with hypermobility such as the Marfan syndrome, Osteogenesis Imperfecta or other types of EDS.
* Co-morbidity with neurological disorders

Inclusion criteria for the control group:

* Able to read and understand Swedish
* Healthy
* Pain free at time of investigation (Numerical Rating Scale score <3/10).

Exclusion criteria for the control group:

* Pregnancy and one year postpartum.
* Past or present signs of rheumatic, neurologic, musculoskeletal, metabolic diseases.
* Chronic pain.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Adolecents diagnosed with HSD/hEDS, at Children's Primary Health Care Clinics in Gothenburg and Southern Bohuslän, and at Queen Silvia Children's Hospital and Skaraborgs hospital Skövde will be asked to participate. In addition, a control group of healthy pain free adolecents, matched for sex, age will be recruited from different schools in the region, throw hospital stuff and social media.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-11-25 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Pressure Pain thresholds, primary and secondary hyperalgesia | Baseline, pre-intervention
  A hand-held pressure algometer (Wagner Instruments, FPX 25) will be used to assess pressure pain thresholds (PPT).
  The 1 cm2 rubber tip of the algometer will be positioned at an angle of 90 degrees in relation to the body part evaluated and pressure will be applied at a rate of 1 kg/s.
  PPT measurements will be carried out on the lower back in the supine position, on the tibialis anterior in the prone position, on the trapezius and deltoid while sitting.
  The participants will be instructed to say "stop" as soon as the sensation of a pressure changes to an uncomfortable feeling. The pressure algometer will be removed immediately and the recorded value will be noted.
  This procedure will be repeated time three times at each test location (30 seconds between each measurement). Average value of the last two measurements is used as the baseline.
  The order of the PPT measurement points will be randomized for each group.
Change of Pressure Pain thresholds, exercise-induced hyperalgesia | Immediately after the intervention
  Exercise-induced hyperalgesia will be measured by repeating the pressure pain thresholds (PPT) measures at the trapezius muscle and the tibialis anterior muscle (as described above) immediately after the performance of an submax exercise test on a bicycle ergometer
  The order of the PPT measurement points in the exercise-induced hyperalgesia measurements will be randomized for each group.

SECONDARY OUTCOMES:
Numerical rating scale | Baseline, pre-intervention and immediately after the intervention
  Average pain intensity will be measured using a 0-10 numerical rating scale (NRS) , with 0 = "no pain" and 10 = "worst possible pain" as the endpoint.
Heart rate | Immediately after the intervention
  Peak heart rate immediately after a cycling test (heartbeat/min) will be recorded.
Borg Rating of Perceived Exertion Scale | Immediately after the intervention
  The subjective perceived effort of physical activity is measured with Borg Rating of Perceived Exertion Scale (Borg's RPE scale).
  Borg´s RPE measures physical activity intensity. Perceived exertion of how hard the individual feels the body is working. The individual experienced physical sensations during physical activity (increased heart rate, increased breathing or breathing rate, increased sweating and muscle fatigue)
  The scale goes from 6 "No effort at all" to 20 "Maximum effort" .
Medical examination | Baseline, pre-intervention
  Medical examination according to the 2017 criteria for Hypermobility Spectrum Disorder or HSD/hEDS (hEDS Diagnostic Checklist).
  Include assessment of joint mobility according to the Beighton scale (described below), physical examination of the diagnostic criteria for hEDS, family history of hEDS, and presence of musculoskeletal pain and joint dislocations.
Beighton scale | Baseline, pre-intervention
  The Beighton scale assesses 9 joints for hypermobility. Hyperextension in elbow joint bilaterally >10 degrees, hyperextension in knee joint bilaterally > 10 degrees, hyperextension of the fifth finger bilaterally > 90 degrees, ability to move the thumb towards the forearm bilaterally and trunk flexion in standing (palm completely on the surface).
  A total of 9 points is possible, generally hypermobility is achieved at 6 points for children and adolescence.
Demographics child | Baseline, pre-intervention
  Back ground data like age, sex ,onset, diagnosis, date of diagnosis, HSD/hED, family history of hypermobility, pain, physical activity habits, the impact of pain on school attendance, and other chronic diseases will be collected through a questionnaire.
  The questionnaire consists of 14 questions, of which 11 are multiple-choice questions, two with numerical rating scale answer options and one pain drawing.
Demographics caregiver | Baseline, pre-intervention
  Back ground data of the caregiver concerning education, type of employment and marital status, family history of pain, the caregiver's experience of the child's pain and physical activity level will be collected through a questionnaire.
  The questionnaire consists of 16 questions, of which 15 are multiple-choice questions, and one pain drawing.
Functional Disability Inventory | Immediately after the intervention
  Functional Disability Inventory (FDI) is a self-report inventory consisting of 15 items that are graded on a five-point scale, ranging from 0 to 4 ("No Trouble" to "Impossible"). The FDI assessed difficulties with the performance of daily activities in home, school, recreational, and social domains. Participants are asked to rate how much difficulty they had completing various tasks, "in the past few days". The sum of answers creates a total score (range 0-60) with higher scores indicating greater pain-related disability. The FDI was created for use in children and adolescents 8-17 years old with recurrent abdominal pain.
Frequency of Participation Questionnaire | Immediately after the intervention
  Participation will be measured using the Frequency of Participation Questionnaire (FPQ). The question is developed to measure the child's participation in all areas of the International Classification of Functioning, Disability and Health.
  FPQ consists of 14 questions about participation in everyday activities such as school and leisure.
  Participants indicate how often an activity is carried out. Grading from 0 ("never") to 5 ("a few times per week").
Multidimensional Fatigue Scale | Immediately after the intervention
  Fatigue will be measured with the Pediatric Quality of Life Inventory (PedsQL) Multidimensional Fatigue Scale.
  PedsQL Multidimensional Fatigue Scale is a self-assessment form that consists of 18 statements that are graded on a five-point scale, from 0 "never a problem" to 4 "almost always a problem". The PedsQL scale consists of three subscales: General Fatigue, Sleep/Rest Fatigue, and Cognitive Fatigue. The Child/Adolescents questionnaire includes ages, 5-7, 8-12 and 13-18.
  Items are reversed scored and linearly transformed to a 0-100 scale, so that higher scores indicate better outcome. To reverse score, the 0-4 scale items will be transformed to 0-100 as follows: 0=100, 1=75, 2=50, 3=25, 4=0.
Pain Catastrophizing scale | Immediately after the intervention
  Catastrophizing will be measured with the child version of the Pain Catastrophizing scale (PCS-C).
  The PCS-C is a self-assessment form that consists of 13 statements that are graded on a five-point scale, from 0 "not at all" to 4 "very much". The total score is 52 points where higher scores indicate higher catastrophizing thoughts. In agreement with previous study using PCS - C to investigate movement loss in children and their parents shared the result on PCS-C in this study into low (0-14 points), between.(15-25 points) and high (26-52) estimated disaster thoughts.
Hospital anxiety and depression scale | Immediately after the intervention
  Anxiety and depression will be measured with the Hospital anxiety and depression scale (HADS).
  HADS is a self-assessment form developed to measure anxiety and depression in patients in somatic care. HADS consists of 14 statements with seven statements for each subscale: HADS anxiety and HADS depression that are graded on a four-point scale from 0 to 3 points. The participant should decide how often he or she has known in the last week, for example "as if something terrible will happen" or whether he or she "appreciates the same things as before". The scores from the seven different statements per sub-scale are combined and can amount to a maximum of 21 points per sub-scale. 0-7 points: Does not speak for anxiety/depression, 8-10 points: The score may be an indication of an anxiety or depression condition in the person, 11 points or more: Demonstrate a likely depression or anxiety of clinical significance.
Physical activity | Continuous measurement over seven days, immediately after the intervention
  Physical activity was measured with Axivity AX3 triaxial accelerometer (Axivity Ltd, UK).
  The participants were instructed to wear it attached to the right thigh with medical tape for seven days.
Diary | Continuous measurement over seven days, immediately after the intervention
  Participants will record planned physical activity and the time when they go to bed and get up parallel to the activity measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Mari Lundberg, Professor, Study Director — University of Gothenborg
Locations (2):
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg, Region Västra Götaland
  - Skaraborgs Hospital Skövde, Skövde, Region Västra Götaland

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Castori M, Tinkle B, Levy H, Grahame R, Malfait F, Hakim A. A framework for the classification of joint hypermobility and related conditions. Am J Med Genet C Semin Med Genet. 2017 Mar;175(1):148-157. doi: 10.1002/ajmg.c.31539. Epub 2017 Feb 1. PMID 28145606
- [Derived] Schubert-Hjalmarsson E, Fridolfsson J, Arvidsson D, Borjesson M, Lundberg M. Exploring physical activity patterns in adolescents with hypermobility spectrum disorder or hypermobile Ehlers-Danlos Syndrome. Pediatr Rheumatol Online J. 2025 Jul 8;23(1):69. doi: 10.1186/s12969-025-01124-0. PMID 40629345
- See also: hEDS Diagnostic Checklist — https://www.ehlers-danlos.com/heds-diagnostic-checklist/